CLINICAL TRIAL: NCT03680339
Title: The Effect of Preoperative and Post Operative Misoprostol Administration on Intraoperative Blood Loss and Postpartum Hemorrhage in CS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 42
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Cesarean Section; Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine ecbolic group (Active Comparator): 100 patients will receive routine ecbolics ( oxytocin) after delivery of baby
  Interventions: Procedure: cesarean section; Drug: Oxytocin
- Misoprostol group (Active Comparator): The 100 patients will receive routine ecbolics (oxytocin) after delivery of baby plus 400 microgram misoprostol rectally with catheterization and another 400 microgram rectally after closure of abdomen
  Interventions: Procedure: cesarean section; Drug: Misoprostol; Drug: Oxytocin

INTERVENTIONS:
Procedure: cesarean section — CS will be done by pfannenstiel incision , transverse lower uterine segment incision ,immediate cord clamping after delivery of baby , closure of uterus by 2 layers , closure of abdomen in layers
Drug: Misoprostol — The 100 patients will receive routine ecbolics (for example oxytocin) after delivery of baby plus 400 microgram misoprostol rectally with catheterization and another 400 microgram rectally after closure of abdomen
  Other Names: Cytotec
  Arms: Misoprostol group
Drug: Oxytocin — 10 IU of oxytocin with fetal delivery

SUMMARY:
• Patients will be divided into two groups 100 patients will receive routine ecbolics (for example oxytocin) after delivery of baby The 100 patients will receive routine ecbolics (for example oxytocin) after delivery of baby plus 400 microgram misoprostol rectally with catheterization and another 400 microgram rectally after closure of abdomen

Then we will compare between two groups regarding

* Intaoperative blood loss
* Risk of Postpartum hemorraghe in the first 24 hrs
* HB pre and postoperative for all patients

Intraoperative blood loss will be estimated by the number and weight of soaked towels and amount of blood in suction unit

DETAILED DESCRIPTION:
• Patients will be divided into two groups 100 patients will receive routine ecbolics (for example oxytocin) after delivery of baby The 100 patients will receive routine ecbolics (for example oxytocin) after delivery of baby plus 400 microgram misoprostol rectally with catheterization and another 400 microgram rectally after closure of abdomen

Then we will compare between two groups regarding

* Intaoperative blood loss
* Risk of Postpartum hemorraghe in the first 24 hrs
* HB pre and postoperative for all patients

Intraoperative blood loss will be estimated by the number and weight of soaked towels and amount of blood in suction unit

ELIGIBILITY:
Inclusion Criteria:

women attending for elective CS.

* Age between 20-35 years.
* Normal placental site
* Normal coagulation profile
* Full term pregnancies(above 37 wks)
* Medically free
* Spinal anesthesia
* Living baby
* Average liquor by U/S

Exclusion Criteria:

* • Women attending for emergency CS

  * .age below 20 or above 35
  * Abnormal placentation (Placenta previa,accrete,increta or percreta)
  * Women with coagulopathy
  * Preterm pregnancies (before 37 wks)
  * Medical disorder (Hypertension,Diabetes, Endocrinal disorder)
  * General anathesia
  * IUFD
  * Oligo or polyhydraminos by U/S

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
postpartum hemorrhage | 24 hours after cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Fawzi T, Shalaby MA, Samy A, Rabee MA, Ali AS, Hussein EA, Hammad B, Deeb WS. A randomized controlled trial of the safety and efficacy of preoperative rectal misoprostol for prevention of intraoperative and postoperative blood loss at elective cesarean delivery. Int J Gynaecol Obstet. 2019 Oct;147(1):102-107. doi: 10.1002/ijgo.12922. Epub 2019 Jul 25. PMID 31304593